CLINICAL TRIAL: NCT05936944
Title: Ruolo Della Luce Naturale Nella Prevenzione Del Delirium Dopo Cardiochirurgia: Studio Osservazionale Prospettico Con Controllo Storico
Brief Title: Role of Natural Light in the Prevention of Delirium After Cardiac Surgery: a Prospective Observational Study With Historical Control
Acronym: iWOnDer
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Davide Nicolotti, Principal Investigator, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: SIRER 6097
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Intensive Care Unit Delirium; Postoperative Delirium; Cardiac Surgery
Keywords: cardiac surgery; postoperative delirium; natural light
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural Light: Group of patients enrolled in the first ICU, with natural lighting
- Artificial Light: Group of patients enrolled in the second ICU, with totally artificial lighting
  Interventions: Other: Exposure to totally artificial lighting

INTERVENTIONS:
Other: Exposure to totally artificial lighting — The second group of patients will be admitted to an ICU without windows and with a totally artificial lighting
  Groups: Artificial Light

SUMMARY:
Postoperative delirium is a common complication that usually occurs acutely within the first 24 hours after surgery and resolves within 72 hours; it is common in all medical areas and particularly affects patients over the age of 65 and those with pre-existing cognitive impairments. It is characterized by difficulty organizing and coordinating thoughts and by slowing down motor functions that are observed for a short period after surgery.

The study will be an observational prospective study with historical control (pre/post-study) whose primary objective is to identify the incidence of postoperative delirium in patients undergoing cardiac surgery. The population will be adult patients undergoing cardiac surgery at our University Hospital over a period of 12 months. The intervention will be exposure to totally artificial light (for patients hospitalized after the relocation of the department to its original location). The comparator will be exposure to natural light (for patients who will be hospitalized during our temporary transfer to an environment with natural lighting). The outcome will be the incidence of delirium, measured with the Confusion Assessment Method-Intensive Care Unit (CAM-ICU) scale; episodes of agitation requiring sedative drugs; time elapsed before onset of delirium. The study will last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* planned cardiac surgery
* planned ICU admission after surgery

Exclusion Criteria:

* cardiac surgery with total suspension of cerebral perfusion
* patient with diagnosed dementia or major depressive disorder
* patient unable to perform CAM-ICU evaluation
* emergent surgery
* patient in ICU before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing cardiac surgery with planned postoperative ICU admission. All tipes of cardiac surgery, irrespective of surgical access or technique, but excluding surgery performed under total circulatory arrest (totale suspension of brain perfusion). Patients will be excluded if they are unable to perform CAM-ICU assessment, if they were diagnosed with major depression or moderate/severe dementia and if they were already in ICU before surgery. Emergent surgery will also be an exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | first five postoperative days or ICU discharge (wichever comes first)
  Occurrence of delirium, diagnosed with at least one positive CAM-ICU evaluation

SECONDARY OUTCOMES:
Postoperative episodes of agitation | first five postoperative days or ICU discharge (wichever comes first)
  number of episodes of postoperative agitation (RASS>+1) requiring farmacological treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Maggiore di Parma, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: Undecided